## Official title:

Assessing the impact of integrative medicine on anxiety and wellbeing of hospital workers exposed directly or indirectly to terror, trauma or war

NCT number: not yet available

Document date: December 20th, 2023

## Background:

In Israel, one of the world's leading treatment concepts has been developed on the subject of mental treatment for trauma as a result of terrorism and war, based on experience in Israel and the world, including in disaster-stricken areas [1]. The incidence and intensity of the trauma that patients and staff members experience depends on many variables, and can involve both those who were directly exposed to the trauma and those who were indirectly exposed (for example: treatment of patients who were exposed to trauma or emotional distress in the general public as a result of a national trauma) [2]. Typical ASD symptoms include hyperarousal; Avoidance (convergence in), dissociation (detachment) and intrusion ("flashbacks") [3]. In these situations, conversational therapy, psychotherapy and other approaches are accepted which are limited in terms of effectiveness in reducing the symptoms and preventing the risk of developing PTSD. Hence the need for additional treatment approaches, such as a combination of treatment with complementary/integrated (integrative) medicine focused on responding to physical distress and reducing arousal more [4].

During the "Iron Swords" war, the residents of the Gaza Strip and the surrounding area, along with the soldiers of the security service, were exposed to a very high intensity of trauma. Added to this is an extensive cycle of trauma for those who were directly and indirectly exposed to loss and terror throughout the country. Medical teams in the hospitals and in the community were exposed with the highest intensity to these traumatic aspects which were amplified by the collapse of many of the resilience and mental health centers in the south.

An integrative medicine treatment clinic was established at the Bnei Zion Medical Center for the purpose of providing a response to all hospital employees who are exposed and will be exposed (directly or indirectly) to the wounded and patients expressing trauma, including symptoms of acute stress disorder, as a result of war and terrorism. Hospital employees are invited to register for complementary medicine treatments on the hospital's website according to indications that include anxiety, emotional distress and/or typical Acute Stress Disorder (ASD) symptoms, including physical distress (such as pain, breathing disorder, digestive system symptoms, exhaustion, etc.). The employees are treated by a team from the system for integrated (integrative) medicine, including practitioners of acupuncture (acupuncture); touch/movement techniques (for example, qigong, reflexology, shiatsu) or mind-body medicine (for example, relaxation and breathing exercises) and may include one or more of the above 3 treatment areas.

In the proposed study, we plan to examine the effect of these treatments on various symptoms experienced by hospital employees during this period.

## Aim:

The purpose of the study is to characterize the hardships of the employees of the Bnei Zion Medical Center in order to evaluate the effect of integrative medicine treatments that can be alleviated on the main hardships, including in the spectrum of acute stress disorder, expressed by the employees whether as a result of direct or indirect exposure to war/terror events and/or as a result of the treatment of casualties.

## Methods:

This is a questionnaire study examining the effect of integrative medicine treatments that are routinely given in a clinic established for all employees of the Bnei Zion Medical Center. The research focuses on the plight of all Bnei Zion Hospital employees, including staff members in the emergency medicine departments, operating room, hospitalization and clinics who are exposed to war/terrorist events and/or as a result of the treatment of casualties.

Evaluation of the research results will be based on the MYCAW - Measure Yourself Concerns and Wellbeing questionnaire. This questionnaire assesses before the start of the integrative intervention the two main distresses that the study participant expects to improve following the integrative treatment, and assesses their severity on a VAS (Visual Analogue Score) scale ranging from 0 to 6. Another question measuring the hospital employee's performance at work on the VAS scale was added to the original MYCAW questionnaire. Another assessment of the MYCAW questionnaire will be carried out 24 hours after the integrative treatment of phone call findings. In addition, a valid questionnaire will be sent that assesses anxiety and mental distress ASD (Acute Stress Disorder) before the start of the treatment and approximately 4-8 weeks later.

The study will be conducted within the Bnai Zion Medical Center during the current emergency. The state of the study will include up to 500 participants and repeat treatments will be possible for the entire hospital staff.

Inclusion criteria: All hospital employees expressing anxiety, emotional distress and/or typical ASD symptoms, including physical distress resulting directly or indirectly from exposure to the trauma of terrorism or war, who receive integrated medical treatments as part of the staff clinic established in Bnei Zion.

Exclusion criteria: none

Conditions for stopping the medical experiment: Staff members who express a desire to stop their participation in the study.

Data analysis:

The data analysis will be conducted using a research methodology that combines quantitative and qualitative aspects. The results of the study and demographic characteristics will be coded in an EXCEL sheet and then into the SPSS software. Descriptive data of the various variables will be produced. The findings will be analyzed with the help of t-test for unpaired tests for prevalence percentages. If necessary, non-parametric tests will be used to compare subpopulations.

Ethical issues of the experiment:

The extraction of the demographic information and its analysis will be done by the researchers. Research data will be coded in an electronic file in a way that will not allow identification of the participants. The study has been approved by the Ethical Committee of Bnai Zion Medical Center (ID: 0105-23-BNZ).

References:

1. Lahad M, Leykin D. Ongoing exposure versus intense periodic exposure to military conflict and terror attacks in Israel. J Trauma Stress. 2010 Dec;23(6):691-8.

2. Koren D, Caspi Y, Leiba R, Bloch D, Vexler B, Klein E. Acute stress reactions among medical and non-medical personnel in a general hospital under missile attacks. Depression Anxiety. 2009;26(2):123-8.

- 3. Lawyer SR, Resnick HS, Galea S, Ahern J, Kilpatrick DG, Vlahov D. Predictors of peritraumatic reactions and PTSD following the September 11th terrorist attacks. Psychiatry. 2006 Summer;69(2):130-41.
- 4. Tan L, Strudwick J, Deady M, Bryant R, Harvey SB. Mind-body exercise interventions for prevention of post-traumatic stress disorder in trauma-exposed populations: a systematic review and meta-analysis. BMJ Open. 2023 Jul 12;13(7):e064758.